CLINICAL TRIAL: NCT04533451
Title: Older Non-Small Cell Lung Cancer Patients (>/= 70 Years of Age) Treated With First-Line MK-3475 (Pembrolizumab)+/- Chemotherapy (Oncologist's/Patient's Choice)
Brief Title: Testing the Effects of MK-3475 (Pembrolizumab) With or Without the Usual Chemotherapy Treatment for Patients 70 Years of Age and Older With Advanced Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A171901; NCI-2020-00544 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH)
Record Dates: First submitted 2020-08-19; First posted 2020-08-31 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Lung Adenocarcinoma; Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Adenocarcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab; Pemetrexed; Carboplatin; Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pembrolizumab; Other: Comprehensive Geriatric Assessment; Other: Questionnaire Administration; Other: Quality-of-Life Assessment
- Group B (pembrolizumab, pemetrexed, carboplatin) (Experimental): Patients receive pembrolizumab IV over 30 minutes, pemetrexed IV over 10 minutes, and carboplatin IV per institutional guidelines on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Other: Comprehensive Geriatric Assessment; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Pembrolizumab — Given IV
Drug: Pemetrexed — Given IV
  Arms: Group B (pembrolizumab, pemetrexed, carboplatin)
Drug: Carboplatin — Given IV
  Arms: Group B (pembrolizumab, pemetrexed, carboplatin)
Other: Comprehensive Geriatric Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This trial studies the side effects of pembrolizumab with or without chemotherapy in treating patients with stage IV non-small cell lung cancer that has come back (recurrent) and has spread to other places in the body (advanced). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as pemetrexed and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab with or without chemotherapy may shrink the tumor in older patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVE:

I. To estimate the adverse event profile of MK-3475 (pembrolizumab) in non-small cell lung cancer patients who are age 70 years of age or older and who are treated with MK-3475 (pembrolizumab) +/- chemotherapy in a first-line setting.

SECONDARY OBJECTIVES:

I. To estimate overall survival. II. To describe patient quality of life during the treatment using the Linear Analogue Self-Assessment (LASA) questionnaire.

III. To explore whether Comprehensive Geriatric Assessment (CGA) -derived risk score is able to predict rates of severe adverse events in older cancer patients who receive MK-3475 (pembrolizumab) or MK-3475 (pembrolizumab) + chemotherapy.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP A: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

GROUP B: Patients receive pembrolizumab IV over 30 minutes, pemetrexed IV over 10 minutes, and carboplatin IV per institutional guidelines on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up annually for up to 5 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of Disease: Histologic or cytologic diagnosis of non-small cell lung cancer (adenocarcinoma). Stage IV or recurrent metastatic non-small cell lung cancer. No planned initiation of definitive (potentially curative) concurrent chemo-radiation
* Planning to begin MK-3475 (pembrolizumab) treatment within 14 days of registration, with or without combination chemotherapy. Treating physician considers pembrolizumab as appropriate and plans to proceed with one of the following treatment schedules:

  * MK-3475 (pembrolizumab) 200 mg IV flat dose every 21 days or 400 mg IV every 42 days.
  * MK-3475 (pembrolizumab) 200 mg IV or 400 mg IV + carboplatin area under the curve (AUC) = 5 + pemetrexed 500 mg/m^2 (20% chemotherapy dose reduction is permitted per the discretion of the treating physician)
* Patients will be ineligible if they have an autoimmune disorder, are post-organ transplantation, or are receiving ongoing immunosuppression treatment
* Prior adjuvant therapy is allowed and must have been completed at least 6 months prior to registration
* No planned radiation or other cancer treatment in the 3 months following registration
* No untreated brain metastases. Patients must be off corticosteroids and asymptomatic at registration
* Absolute neutrophil count (ANC) >= 1500/mm^3 (1.5 x 10^9/L)
* Platelet count: >= 100,000/mm^3 (100 x 10^9/L)
* Creatinine >= 30 mL/min* for patients enrolled to pembrolizumab alone and > 45 mL/min for patients enrolled to chemotherapy + pembrolizumab

  * Calculated using the Cockcroft-Gault formula
* Total serum bilirubin =< 1.5 upper limit of normal (ULN) (< 3 ULN if Gilbert's disease)
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 3 x ULN (=< 5.0 x ULN if liver metastases present)
* Alkaline phosphatase =< 2.5 x ULN (=< 5 x ULN if bone or liver metastases present) Language: Patients must be able to speak and comprehend English in order to complete the mandatory patient-completed measures

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2027-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (505):
- United States (505):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Saint Helena Hospital, St. Helena, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Morton Plant Hospital, Clearwater, Florida
  - South Florida Baptist Hospital, Plant City, Florida
  - Saint Anthony's Hospital Cancer Care Center, St. Petersburg, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Jennie Edmundson Memorial Hospital, Council Bluffs, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner LSU Health Saint Mary's Medical Center, Shreveport, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Veteran's Affairs Medical Center - Saint Louis, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - South Nassau Cancer Center, Valley Stream, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Johnston Health Clayton, Clayton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kenansville, Kenansville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Scotland Memorial Hospital-Laurinburg Cancer Center, Laurinburg, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Vidant Oncology-Richlands, Richlands, North Carolina
  - Johnston Memorial Hospital, Smithfield, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Zangmeister Center Grove City, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Good Samaritan Hospital, Corvallis, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Kent Hospital, Warwick, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Cancer Specialists of Tidewater Limited, Chesapeake, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Westchester Emergency Center, Midlothian, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Riverside Shore Cancer Center, Onancock, Virginia
  - Bon Secours Maryview Medical Center, Portsmouth, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - Cancer Specialists of Tidewater-Suffolk, Suffolk, Virginia
  - Peninsula Cancer Institute-Cancer Specialists of Tidewater, Virginia Beach, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (Pembrolizumab): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.>> >> Pembrolizumab: Given IV>>
  >> Comprehensive Geriatric Assessment: Ancillary studies>>
  >> Questionnaire Administration: Ancillary studies>>
  >> Quality-of-Life Assessment: Ancillary studies
- Group B (Pembrolizumab, Pemetrexed, Carboplatin): Patients receive pembrolizumab IV over 30 minutes, pemetrexed IV over 10 minutes, and carboplatin IV per institutional guidelines on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.>> >> Pembrolizumab: Given IV>>
  >> Pemetrexed: Given IV>>
  >> Carboplatin: Given IV>>
  >> Comprehensive Geriatric Assessment: Ancillary studies>>
  >> Questionnaire Administration: Ancillary studies>>
  >> Quality-of-Life Assessment: Ancillary studies
Period: Overall Study
Arm/Group | Group A (Pembrolizumab) | Group B (Pembrolizumab, Pemetrexed, Carboplatin)
Started | 45 | 56
Completed | 43 | 52
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Pembrolizumab) | Group B (Pembrolizumab, Pemetrexed, Carboplatin) | Total
Number analyzed (Participants) | 45 | 56 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.0 (5.85) | 76.1 (4.21) | 77.8 (5.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 20 | 33 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 43 | 53 | 96
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 37 | 45 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 5
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction.> ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.> ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.> ECOG = 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours.> ECOG = 0 is better. ECOG = 3 is worse.
  Participants
    0 | 11 | 21 | 32
    1 | 25 | 32 | 57
    2 | 9 | 2 | 11
    3 | 0 | 1 | 1
Concomitant Chemo [Count of Participants; unit: Participants]
  No | 45 | 15 | 60
  Yes | 0 | 41 | 41
Prior Adjuvant Chemo [Count of Participants; unit: Participants]
  No | 40 | 52 | 92
  Yes | 5 | 4 | 9
Prior Radiotherapy [Count of Participants; unit: Participants]
  No | 34 | 42 | 76
  Yes | 11 | 14 | 25
Any Prior Cancer Diagnosed [Count of Participants; unit: Participants]
  No | 34 | 39 | 73
  Yes | 11 | 17 | 28
Cancer Treatment started prior to enrollment [Count of Participants; unit: Participants]
  No | 39 | 50 | 89
  Yes | 6 | 6 | 12
Smoking History [Count of Participants; unit: Participants]
  No | 3 | 3 | 6
  Yes | 42 | 53 | 95
PD-L1 Expression [Mean (Standard Deviation); unit: Tumor Proportion Score (%)] | 54.1 (37.35) | 13.6 (25.84) | 32.1 (37.43)
Diagnosis of Non-Small Cell Lung Cancer [Count of Participants; unit: Participants]
  Recurrent Metastatic | 6 | 9 | 15
  Stage IV | 39 | 47 | 86

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade 3 or Worse Adverse Events Post Registration
Description: Assessed by National Cancer Institute Common Terminology Criteria in Adverse Events version 5.0. The proportion of patients experience grade 3 or worse adverse events (AEs) will be summarized by frequency and percentage along with a 95% confidence interval (CI) separately by type of therapy (monotherapy or combination therapy) as well as combining the two cohorts. All other individual AEs will be analyzed in an exploratory and hypothesis generating manner; including and not limited to multi-variate logistic regression models considering the baseline demographics and the presence/absence of the AE.
Time Frame: Up to 7 days of last day of treatment, up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Group A (Pembrolizumab): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.> >>
  >
  >> Pembrolizumab: Given IV>
  >>
  >
  >> Comprehensive Geriatric Assessment: Ancillary studies>
  >>
  >
  >> Questionnaire Administration: Ancillary studies>
  >>
  >
  >> Quality-of-Life Assessment: Ancillary studies
- Group B (Pembrolizumab, Pemetrexed, Carboplatin): Patients receive pembrolizumab IV over 30 minutes, pemetrexed IV over 10 minutes, and carboplatin IV per institutional guidelines on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.> >>
  >
  >> Pembrolizumab: Given IV>
  >>
  >
  >> Pemetrexed: Given IV>
  >>
  >
  >> Carboplatin: Given IV>
  >>
  >
  >> Comprehensive Geriatric Assessment: Ancillary studies>
  >>
  >
  >> Questionnaire Administration: Ancillary studies>
  >>
  >
  >> Quality-of-Life Assessment: Ancillary studies
Arm/Group | Group A (Pembrolizumab) | Group B (Pembrolizumab, Pemetrexed, Carboplatin)
Number analyzed (Participants) | 43 | 52
Participants | 11 | 22

2. Secondary Outcome: Overall Survival (OS)
Description: Will be summarized using the Kaplan-Meier estimator, separately by monotherapy or combination therapy as well as by the combined cohort.
Time Frame: From study registration to death or the last follow-up whichever occurs first, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A (Pembrolizumab) | Group B (Pembrolizumab, Pemetrexed, Carboplatin)
Number analyzed (Participants) | 43 | 52
months | 16.4 [10.1 to NA] — Not enough events after median | 29.9 [16.4 to NA] — Not enough events after median
Statistical Analysis 1: Comparison: Group A (Pembrolizumab) vs Group B (Pembrolizumab, Pemetrexed, Carboplatin); Test type: Superiority; p = 0.0385, Log Rank

3. Secondary Outcome: Quality of Life (QOL): Linear Analogue Self-Assessment [LASA] Questionnaire
Description: The overall quality of life score (the first question of the Linear Analogue Self-Assessment [LASA] questionnaire) at each time point as well as change from baseline will be summarized by mean (standard deviation), median (range) along with a longitudinal plot. The median quality of life (QOL) change from baseline along with a 95% confidence interval (CI) will be estimated using the Hodges-Lehmann method. The overall quality of life score will be measured on a scale from 0-10, with higher being better.
Time Frame: Up to 9 weeks
Population: There were 60 patients who had QOL change from baseline to week 9. Per the protocol section 13.5, quality of life would be examined combined by arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Combined Arms: Arms A and arms B
Arm/Group | Combined Arms
Number analyzed (Participants) | 60
score on a scale | 0.0 [-1 to 1]

4. Secondary Outcome: Comprehensive Geriatric Assessment Risk Score
Description: The geriatric risk score, measured as low, medium, or high, will be summarized in a 3X2 frequency table with adverse events.
Time Frame: At baseline. Per the protocol section 13.5,Comprehensive geriatric assessment would be examined combined by arm.
Population: Analyzed with both arms combined
Measure: Count of Participants; unit: Participants
Groups:
- Combined Group: Patients from both Arms A and arms B
Arm/Group | Combined Group
Number analyzed (Participants) | 95
Participants
  Low Risk Group | 14
  Medium Risk Group | 15
  High Risk Group | 4
Statistical Analysis 1: Comparison: Combined Group; Test type: Equivalence — Relatively large sample size and groups are independent; p = 0.9829, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Group A (Pembrolizumab) | Group B (Pembrolizumab, Pemetrexed, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 8/43 | 6/54
Serious Adverse Events (participants affected / at risk) | 8/43 | 6/54
Other Adverse Events (participants affected / at risk) | 43/43 | 53/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Pembrolizumab) (N=43) | Group B (Pembrolizumab, Pemetrexed, Carboplatin) (N=54)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 5 (5) | 5 (5)
Disease progression (General disorders) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Pembrolizumab) (N=43) | Group B (Pembrolizumab, Pemetrexed, Carboplatin) (N=54)
Anemia (Blood and lymphatic system disorders) | 23 (173) | 46 (338)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (17) | 1 (39)
Eosinophilia (Blood and lymphatic system disorders) | 2 (3) | 2 (13)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 4 (4)
Chest pain - cardiac (Cardiac disorders) | 1 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (12)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 2 (31) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (12) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 3 (8)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 7 (87) | 15 (71)
Blurred vision (Eye disorders) | 5 (24) | 2 (2)
Cataract (Eye disorders) | 1 (14) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 2 (2)
Flashing lights (Eye disorders) | 1 (6) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 11 (22) | 13 (23)
Belching (Gastrointestinal disorders) | 1 (20) | 1 (2)
Constipation (Gastrointestinal disorders) | 14 (94) | 29 (175)
Diarrhea (Gastrointestinal disorders) | 14 (35) | 24 (58)
Dry mouth (Gastrointestinal disorders) | 3 (12) | 3 (14)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (4) | 1 (3)
Dysphagia (Gastrointestinal disorders) | 1 (6) | 2 (9)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (19) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (3) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 4 (7)
Nausea (Gastrointestinal disorders) | 14 (31) | 35 (109)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (14) | 11 (13)
Chills (General disorders) | 1 (2) | 1 (6)
Edema face (General disorders) | 1 (9) | 0 (0)
Edema limbs (General disorders) | 4 (22) | 5 (30)
Facial pain (General disorders) | 0 (0) | 1 (4)
Fatigue (General disorders) | 33 (215) | 50 (376)
Fever (General disorders) | 0 (0) | 5 (5)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (2) | 1 (3)
Generalized edema (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (17) | 2 (2)
Pain (General disorders) | 4 (17) | 4 (12)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 2 (3)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 1 (3) | 2 (2)
Lung infection (Infections and infestations) | 4 (5) | 4 (5)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (7) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 0 (0) | 4 (4)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (3)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (4)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (6)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (5) | 16 (47)
Alkaline phosphatase increased (Investigations) | 6 (12) | 12 (44)
Aspartate aminotransferase increased (Investigations) | 7 (8) | 9 (21)
Blood bilirubin increased (Investigations) | 5 (5) | 4 (13)
Blood lactate dehydrogenase increased (Investigations) | 3 (9) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 7 (21) | 8 (22)
Investigations - Other, specify (Investigations) | 2 (23) | 2 (7)
Lymphocyte count decreased (Investigations) | 5 (27) | 18 (65)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 16 (44)
Platelet count decreased (Investigations) | 4 (12) | 19 (50)
Thyroid stimulating hormone increased (Investigations) | 2 (4) | 0 (0)
Weight loss (Investigations) | 7 (18) | 3 (16)
White blood cell decreased (Investigations) | 1 (1) | 14 (24)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 24 (93) | 26 (104)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (56) | 16 (68)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperlipidemia (Metabolism and nutrition disorders) | 2 (5) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (22) | 10 (36)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 4 (9)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 5 (8) | 10 (21)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 6 (14)
Hyponatremia (Metabolism and nutrition disorders) | 5 (31) | 10 (24)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (125) | 13 (70)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (14) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (22) | 7 (28)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (14) | 7 (14)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (6) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (10) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (21) | 1 (6)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 5 (15) | 10 (53)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (5) | 4 (5)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (7) | 9 (23)
Memory impairment (Nervous system disorders) | 1 (2) | 1 (1)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 0 (0)
Muscle weakness right-sided (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (4) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 13 (66) | 12 (80)
Presyncope (Nervous system disorders) | 0 (0) | 2 (3)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (20) | 6 (21)
Confusion (Psychiatric disorders) | 3 (31) | 5 (31)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 3 (6)
Insomnia (Psychiatric disorders) | 8 (12) | 9 (26)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 3 (5) | 1 (7)
Dysuria (painful urination) (Renal and urinary disorders) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 5 (15)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 2 (2)
Vaginal dryness (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (9) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (215) | 36 (207)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 30 (199) | 40 (228)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (23) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (9)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 5 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (12) | 2 (9)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (22) | 2 (2)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 3 (11) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (9) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (15) | 7 (16)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (24) | 9 (10)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (8)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 9 (48) | 11 (51)
Hypotension (Vascular disorders) | 4 (10) | 4 (5)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT04533451/Prot_SAP_000.pdf